CLINICAL TRIAL: NCT00562445
Title: Evaluation of the Incidence and Relevance of the Adrenal Insufficiency in Critical Emergencies in Digestive Diseases (GI Bleeding and Acute Pancreatitis)
Brief Title: Adrenal Insufficiency in Critical Emergencies in Digestive Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Other Study IDs: ISRRA-HDA2007; EudraCT: 2007-002355-16
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Digestive Diseases; Adrenal Insufficiency; Gastrointestinal Bleeding; Variceal Bleeding; Acute Pancreatitis
Keywords: Adrenal insufficiency; GI bleeding; Portal hypertension; Acute pancreatitis; Critical emergencies in digestive diseases; Severe acute pancreatitis
MeSH Terms: conditions — Digestive System Diseases; Adrenal Insufficiency; Gastrointestinal Hemorrhage; Pancreatitis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Peptic bleeding
- 2: Portal hypertension bleeding
- 3: Severe acute pancreatitis

SUMMARY:
Observational study about the incidence of relative adrenal insufficiency in patients with cirrhosis and acute variceal bleeding; in patients with acute peptic gastrointestinal bleeding and without liver disease; and in patients with severe acute pancreatitis.

This is a study using pharmaceutical specialties in the approved conditions of use.

DETAILED DESCRIPTION:
Observational, prospective, open-label, in-patient study, that includes patients with upper gastrointestinal bleeding of variceal or peptic origin, and in patients with severe acute pancreatitis.

The adrenal function of every patient included will be evaluated in the first 24 hours of admission This assessment shall be performed using the corticotropin-stimulation short test (synacthen test), that includes serum and saliva determination of cortisol, in basal conditions and 30 and 60 minutes after the administration of 250 ug of corticotropin synthetic (Synacthen, Novartis Pharma AG, Basel, Switzerland).

The cortisol levels will be determined by competitive immunoassay using direct chemoluminescence technology (Bayer Corporation, Pittsburgh, PA, USA).

In patients with severe acute pancreatitis all of these determinations will be repeated at the third day of admission.

Several other clinical and biochemical features will be recorded.

ELIGIBILITY:
Inclusion Criteria (one of the following):

* Presence of acute upper gastrointestinal bleeding (variceal or peptic) + presence of hypovolemic shock (defined as a systolic blood pressure <100 mmHg coupled with a heart rate> 100 ppm), or Hb < 80 g / L;
* Acute pancreatitis (diagnosed by clinical, radiological and biochemical features)with severity criteria (At least one of the following: index of Ranson > 3, APACHE II > 8 or CPR> 120 mg/L, Balthazar CT grade E)

Exclusion Criteria:

* Age <18 years and >80 years.
* Pregnancy.
* Patient refusal to participate in the study.
* Prior corticosteroids treatment(oral or topical).
* Treatment during the 30 days prior to inclusion with any of the following drugs: contraception, etomidate, ketoconazole, rifampin or phenytoin.
* History of cranial trauma or surgery.
* Any malignancy in treatment or progression.
* HIV infection.
* Prior known adrenal pathology.
* Patients not eligible to any active treatment because the existence of any clinical condition considered terminal.
* Patients with associated traumatic blood loss, or any other extraintestinal source of active bleeding.
* Burns.
* Patients who have been previously included in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to our centre that meet inclusion criteria and do not meet exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2007-05; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Relative adrenal insufficiency | 1 week

SECONDARY OUTCOMES:
Therapeutic failure | 45 days
Survival | 45 days
Variations in portal hypertension. | 7 days
Need for vasopressive drugs | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Candid Villanueva, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- HospitalSCSP, Barcelona, Barcelona, Spain